CLINICAL TRIAL: NCT01820208
Title: Efficacy of G-CSF in the Management of Steroid Non-responsive Severe Alcoholic Hepatitis. - A Double Blind Randomized Control Trial.
Brief Title: Efficacy of G-CSF in the Management of Steroid Non-responsive Severe Alcoholic Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS- AH-01
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2016-08

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo would be given s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses)
  Interventions: Drug: G-CSF
- G-CSF (Experimental): G-CSF would be given at a dose of 5 microgram/kg daily for 5 days followed by once in 3 days for a total of 12 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: G-CSF — G-CSF would be given at a dose of 5 microgram/kg daily for 5 days followed by once in 3 days for a total of 12 doses.
  Arms: Placebo
Drug: Placebo — Placebo would be given s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 28 (total 12 doses)
  Arms: G-CSF

SUMMARY:
After successful screening, first the investigators first treat patients of severe alcoholic hepatitis with steroids for 7 days. Patients who are found to be unresponsive as per Lille's score [>0.45] would be randomized into either placebo group or G-CSF group. Responders to steroids will continue on steroids for 28 days followed by 2 weeks of tapering. Non responders will be randomized to receive G-CSF for 28days.

ELIGIBILITY:
Inclusion Criteria:

- Severe alcoholic hepatitis patients [Maddrey's score > 32] aged between 18 to 65 years.

Exclusion Criteria:

* Presence of active infections
* Acute GI bleed
* Hepatorenal syndrome
* Patient unwilling
* DF>120
* Autoimmune hepatitis
* Hepatitis B, Hepatitis C, HIV cases
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Survival of subjects in both group | 4 weeks and 12 weeks

SECONDARY OUTCOMES:
Improvement in Child's score in steroid unresponsive patients with severe alcoholic hepatitis patients | 4 weeks and 12 weeks
  Change in child score at 4 week and 12 weeks compared to baseline in both groups.
Improvement in MELD score in steroid unresponsive patients with severe alcoholic hepatitis patients | 4 weeks and 12 weeks
  Change in MELD score at 4 week and 12 weeks compared to baseline in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Shasthry SM, Sharma MK, Shasthry V, Pande A, Sarin SK. Efficacy of Granulocyte Colony-stimulating Factor in the Management of Steroid-Nonresponsive Severe Alcoholic Hepatitis: A Double-Blind Randomized Controlled Trial. Hepatology. 2019 Sep;70(3):802-811. doi: 10.1002/hep.30516. Epub 2019 Mar 25. PMID 30664267